CLINICAL TRIAL: NCT02636946
Title: A Comparison of Bimatoprost SR to Selective Laser Trabeculoplasty in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-095; 2015-003631-34 (EudraCT Number)
Record Dates: First submitted 2015-12-10; First posted 2015-12-22 (Estimated); Results first posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Glaucoma; Open-Angle Ocular Hypertension
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) (Active Comparator): Primary Eye: Selective Laser Trabeculoplasty (SLT) administered on Day 1 followed by up to three Sham Bimatoprost sustained release (Bim SR) administrations at Day 4 (Cycle 1), Weeks 16 (Cycle 2) and 32 (Cycle 3) or two Sham Bimatoprost SR administrations at Day 4 (Cycle 1) and Week 16 (Cycle 2) for participants who were enrolled under Protocol Amendment 2 or later.
  Contralateral (Other) Eye: Sham SLT administered on Day 1 followed by up to three Bimatoprost SR 15 μg administrations at Day 4 (Cycle 1), Weeks 16 (Cycle 2) and 32 (Cycle 3) or two Bimatoprost SR 15 μg administrations at Day 4 (Cycle 1) and Week 16 (Cycle 2) for participants enrolled under Protocol Amendment 2 or later.
  Interventions: Drug: Bimatoprost SR; Drug: Sham Bimatoprost SR; Procedure: Selective Laser Trabeculoplasty; Procedure: Sham Selective Laser Trabeculoplasty
- Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) (Experimental): Primary Eye: Sham SLT administered on Day 1 followed by up to three Bimatoprost SR 15 μg administrations at Day 4 (Cycle 1), Weeks 16 (Cycle 2) and 32 (Cycle 3) or two Bimatoprost SR 15 μg administrations at Day 4 (Cycle 1) and Week 16 (Cycle 2) for participants who were enrolled under Protocol Amendment 2 or later.
  Contralateral (Other) Eye: SLT administered on Day 1 followed by up to three Sham Bimatoprost SR administrations at Day 4 (Cycle 1), Weeks 16 (Cycle 2) and 32 (Cycle 3) or two Sham Bimatoprost SR administrations at Day 4 (Cycle 1) and Week 16 (Cycle 2) for participants who were enrolled under Protocol Amendment 2 or later.
  Interventions: Drug: Bimatoprost SR; Drug: Sham Bimatoprost SR; Procedure: Selective Laser Trabeculoplasty; Procedure: Sham Selective Laser Trabeculoplasty

INTERVENTIONS:
Drug: Bimatoprost SR — Up to three Bimatoprost SR 15 micrograms (μg) administrations at Day 4, Weeks 16 and 32 (Stage 1) or two Bimatoprost SR 15 μg administrations at Day 4 and Week 16 (Stage 2).
Drug: Sham Bimatoprost SR — Up to three Sham Bimatoprost SR administrations at Day 4, Weeks 16 and 32 (Stage 1) or two Sham Bimatoprost SR administrations at Day 4 and Week 16 (Stage 2).
Procedure: Selective Laser Trabeculoplasty — Selective Laser Trabeculoplasty administered on Day 1.
Procedure: Sham Selective Laser Trabeculoplasty — Sham Selective Laser Trabeculoplasty administered on Day 1.

SUMMARY:
This study will evaluate the intraocular pressure (IOP)-lowering effect and safety of Bimatoprost SR compared with selective laser trabeculoplasty in participants with open-angle glaucoma or ocular hypertension who are not adequately managed with topical IOP-lowering medication for reasons other than medication efficacy (e.g., due to intolerance or nonadherence).

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of either Open-Angle Glaucoma or Ocular Hypertension in each eye that require IOP lowering treatment.

Exclusion Criteria:

* Eye surgery (including cataract surgery) and or eye laser surgery within the past 6 months.
* Enrollment in other studies using Bimatoprost SR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margot Goodkin, Study Director — Allergan
Locations (33):
- United States (21):
  - Eye Center South, Dothan, Alabama
  - Arizona Eye Center, Chandler, Arizona
  - Walman Eye Center, Chandler, Arizona
  - Shasta Eye Medical Group, Inc., Redding, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Eye Associates of Colorado Springs, Colorado Springs, Colorado
  - West Coast Eye Institute, Lecanto, Florida
  - Emory University Eye Center, Atlanta, Georgia
  - Coastal Research Associates, LLC, Roswell, Georgia
  - The Eye Care Institute, Louisville, Kentucky
  - Fraser Eye Center, Fraser, Michigan
  - Galanis Cataract and Laser Eye Center, St Louis, Missouri
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Asheville Eye Associates, Asheville, North Carolina
  - James D. Branch MD, Winston-Salem, North Carolina
  - Bergstrom Eye Research, LLC, Fargo, North Dakota
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - The Cataract & Glaucoma Center, El Paso, Texas
  - DCT- Shah Research, Mission, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Vistar Eye Center, Roanoke, Virginia
- Marsden Eye Specialists, Parramatta, New South Wales, Australia
- Glostrup Hospital, Glostrup Municipality, Capital Region, Denmark
- CHU de Bordeaux Hopital Pellegrin Service Ophtalmologie, Bordeaux, France
- Poland (2):
  - Prywatna Klinika Okulistyczna OFTALMIKA, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Diagnostykii Mikrochirurgii Oka LENS ul., Olsztyn, Warmian-Masurian Voivodeship
- Russia (2):
  - S. Fyodorov Eye Microsurgery Federal State Institution, Novosibirsk Branch, Novosibirsk
  - Ophthalmic Clinical Hospital V.P. Vyhodtseva, Omsk
- Singapore National Eye Centre, Singapore, Singapore
- Spain (2):
  - Centro de Oftalmologia Barraquer, Barcelona
  - Hospital Clinico San Carlos, Madrid
- Thailand (2):
  - Chiang Mai University CMU - Maharaj Nakhon Chiang Mai Hospital, Chiang Mai
  - Thammasat University Hospital, Pathum Thani

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/search-results/?SearchTerm=NCT02636946&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&GenderDescriptions=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&hasResults=&isHighValue=&SortField=&SortOrder=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 144 participants were randomized with 72 participants in each treatment group. Out of them 142 participants were treated. The primary eye was defined as the eye with the higher intraocular pressure (IOP) at Baseline. If both the eyes were the same, the right eye was used as the primary eye. The contralateral eye is the other eye.
Period: Cycle 1 (Day 1 to Week 15)
Arm/Group | SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) | Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye)
Started | 72 | 72
Received Treatment in Either Eye | 72 | 70
Completed | 71 | 67
Not Completed | 1 | 5
Not completed — Withdrawal of Consent | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Reason not Specified | 0 | 1
Not completed — Randomized but not Treated | 0 | 2
Period: Cycle 2 (Week 16 to Week 31)
Arm/Group | SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) | Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye)
Started (Started=received administration (Sham or Bimatoprost SR) in the cycle) | 65 | 62
Completed | 63 | 61
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1
Period: Cycle 3 (Week 32 to Week 52)
Arm/Group | SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) | Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye)
Started (Started=received administration (Sham or Bimatoprost SR) in the cycle) | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population was defined as all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) | Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.2) | 62.1 (11.4) | 60.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 39 | 67
  Male | 44 | 33 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 53 | 59 | 112
  Black or African American | 12 | 9 | 21
  Asian | 5 | 3 | 8
  Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 11 | 7 | 18
  Non-Hispanic | 61 | 64 | 125
  Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) at Baseline
Description: IOP is a measurement of the fluid pressure inside the eye. Measurements were taken at Hour 0.
Time Frame: Baseline (prior to treatment)
Population: Modified Intent-to-Treat (mITT) Population was defined based in the Intent-to-Treat (ITT) population but excluded participants who did not receive the second implant after implementation of Amendment 3.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Groups:
- Selective Laser Trabeculoplasty: SLT administered on Day 1.
  Participants' primary eyes from 'SLT (Primary Eye) / Bim SR 15 ug (Contralateral Eye)' arm and contralateral eyes from 'Bim SR 15 ug (Primary Eye) / SLT (Contralateral Eye)' arm were combined for outcome measure analyses.
- Bim SR 15 μg: Three Bimatoprost SR 15 μg administrations at Day 4 (Cycle 1), Weeks 16 (Cycle 2) and 32 (Cycle 3) or two Bimatoprost SR 15 μg administrations at Day 4 (Cycle 1) and Week 16 (Cycle 2) for participants who were enrolled under Protocol Amendment 2 or later.
  Participants' contralateral eyes from 'SLT (Primary Eye) / Bim SR 15 ug (Contralateral Eye)' arm and primary eyes from 'Bim SR 15 ug (Primary Eye) / SLT (Contralateral Eye)' arm were combined for outcome measure analyses.
Arm/Group | Selective Laser Trabeculoplasty | Bim SR 15 μg
Number analyzed (Participants) | 138 | 138
millimeters of mercury (mmHg) | 24.45 (2.75) | 24.38 (2.49)

2. Primary Outcome: Change From Baseline in IOP at Week 4
Description: IOP is a measurement of the fluid pressure inside the eye. Measurements were taken at Hour 0. A negative change from Baseline indicates an improvement and a positive change from Baseline indicates a worsening. A mixed-effects model with repeated measures (MMRM) was used for analyses.
Time Frame: Baseline (prior to treatment) to Week 4
Population: mITT Population was defined based in the ITT population but excluded participants who did not receive the second implant after implementation of Amendment 3. Overall number analyzed are number of participants and eyes with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Selective Laser Trabeculoplasty | Bim SR 15 μg
Number analyzed (Participants) | 131 | 135
Number analyzed (eyes) | 131 | 135
mmHg | -6.28 (0.30) | -6.98 (0.29)
Statistical Analysis 1: Comparison: Selective Laser Trabeculoplasty vs Bim SR 15 μg; Change from Baseline at Week 4: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to SLT if the upper limit of the 95% CI was ≤ 1.5 mmHg at all scheduled visits (Weeks 4, 12, and 24); Test type: Non-Inferiority — MMRM was used for IOP change from baseline. The model includes IOP change from baseline as the response variable and treatment, visit, eye, baseline IOP, treatment-by-baseline, treatment-by-eye, treatment-by-visit, visit-by-eye interactions as covariates. A Kronecker product of unstructured covariance matrix for study visit and compound symmetry covariance matrix for between eye correlation was used in the analysis; p = 0.0166, MMRM; Least-squares Mean Difference = -0.70, 95% CI 2-sided [-1.28 to -0.13], Standard Error of Mean 0.29

3. Primary Outcome: Change From Baseline in IOP at Week 12
Description: IOP is a measurement of the fluid pressure inside the eye. Measurements were taken at Hour 0. A negative change from Baseline indicates an improvement and a positive change from Baseline indicates a worsening. A MMRM was used for analyses.
Time Frame: Baseline (prior to treatment) to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Selective Laser Trabeculoplasty | Bim SR 15 μg
Number analyzed (Participants) | 122 | 128
Number analyzed (eyes) | 122 | 128
mmHg | -6.28 (0.29) | -6.81 (0.29)
Statistical Analysis 1: Comparison: Selective Laser Trabeculoplasty vs Bim SR 15 μg; Change from Baseline at Week 12: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to SLT if the upper limit of the 95% CI was ≤ 1.5 mmHg at all scheduled visits (Weeks 4, 12, and 24); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.0735, MMRM; Least-squares Mean Difference = -0.52, 95% CI 2-sided [-1.09 to 0.05], Standard Error of Mean 0.29

4. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) at Week 24
Description: as for outcome 3
Time Frame: Baseline (prior to treatment) to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Selective Laser Trabeculoplasty | Bim SR 15 μg
Number analyzed (Participants) | 117 | 126
Number analyzed (eyes) | 117 | 126
mmHg | -6.34 (0.29) | -6.59 (0.29)
Statistical Analysis 1: Comparison: Selective Laser Trabeculoplasty vs Bim SR 15 μg; Change from Baseline at Week 24: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to SLT if the upper limit of the 95% confidence interval (CI) was ≤ 1.5 mmHg at all scheduled visits (Weeks 4, 12, and 24); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.3928, MMRM; Least-squares Mean Difference = -0.25, 95% CI 2-sided [-0.81 to 0.32], Standard Error of Mean 0.29

5. Secondary Outcome: Change From Baseline in IOP at Weeks 8, 15, and 20
Description: IOP is a measurement of the fluid pressure inside the eye. Measurements were taken at Hour 0. A negative change from Baseline indicates an improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (prior to treatment) to Weeks 8, 15 and 20
Population: ITT Population was defined as all randomized participants. Number analyzed is the number of participants and eyes analyzed at the given timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Selective Laser Trabeculoplasty | Bim SR 15 μg
Number analyzed (Participants) | 144 | 144
Number analyzed (eyes) | 144 | 144
mmHg
  Change from Baseline at Week 8: number analyzed (Participants) | 133 | 137
  Change from Baseline at Week 8: number analyzed (eyes) | 133 | 137
  Change from Baseline at Week 8 | -6.65 (3.10) | -7.09 (2.93)
  Change from Baseline at Week 15: number analyzed (Participants) | 126 | 133
  Change from Baseline at Week 15: number analyzed (eyes) | 126 | 133
  Change from Baseline at Week 15 | -6.14 (3.47) | -5.36 (3.73)
  Change from Baseline at Week 20: number analyzed (Participants) | 8 | 7
  Change from Baseline at Week 20: number analyzed (eyes) | 8 | 7
  Change from Baseline at Week 20 | -5.06 (3.33) | -4.29 (1.93)

6. Secondary Outcome: Time to Initial Use of Nonstudy IOP-lowering Treatment as Determined by the Investigator
Description: Median time in days from first treatment to the initial use of non-study IOP-lowering treatment.
Time Frame: First treatment to end of study (up to 525 days)
Population: ITT Population was defined as all randomized participants. Overall number analyzed are number of participants and eyes with data available for analyses.
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: eyes
Arm/Group | Selective Laser Trabeculoplasty | Bim SR 15 μg
Number analyzed (Participants) | 142 | 141
Number analyzed (eyes) | 142 | 141
days | 410 [392.0 to NA] — The upper limit of 95% confidence interval was not estimable due to the low number of participants with events. | 446 [407.0 to NA] — The upper limit of 95% confidence interval was not estimable due to the low number of participants with events.

7. Secondary Outcome: Percentage of Participants With Eyes Achieving a ≥ 20% Reduction in IOP
Description: IOP is a measurement of the fluid pressure inside the eye. Measurements were taken at Hour 0. The participants who did not continue in the subsequent cycle were followed up to Week 52 in Cycle 1, Week 36 in Cycle 2, and Week 20 in Cycle 3.
Time Frame: Baseline (prior to treatment) to Cycle 1: Day 2, Weeks 4, 8, 12, 15, 20, 24, 28, 31, 36, 40, 44, 47, 52; Cycle 2:Day 2, Weeks 4, 8, 12, 15, 20, 24, 28, 31, 36; Cycle 3: Day 2, Weeks 4, 8, 15, 20
Population: ITT Population was defined as all randomized participants. Number analyzed is number of participants and eyes analyzed at the given timepoint.
Measure: Number; unit: percentage of participants
Units Other Than Participants: eyes
Arm/Group | Selective Laser Trabeculoplasty | Bim SR 15 μg
Number analyzed (Participants) | 144 | 144
Number analyzed (eyes) | 144 | 144
percentage of participants
  Cycle 1 Day 2: number analyzed (Participants) | 137 | 137
  Cycle 1 Day 2: number analyzed (eyes) | 137 | 137
  Cycle 1 Day 2 | 60.6 | 92.7
  Cycle 1 Week 4: number analyzed (Participants) | 141 | 141
  Cycle 1 Week 4: number analyzed (eyes) | 141 | 141
  Cycle 1 Week 4 | 70.2 | 78.0
  Cycle 1 Week 8: number analyzed (Participants) | 140 | 140
  Cycle 1 Week 8: number analyzed (eyes) | 140 | 140
  Cycle 1 Week 8 | 72.9 | 80.0
  Cycle 1 Week 12: number analyzed (Participants) | 137 | 137
  Cycle 1 Week 12: number analyzed (eyes) | 137 | 137
  Cycle 1 Week 12 | 67.9 | 75.2
  Cycle 1 Week 15: number analyzed (Participants) | 134 | 134
  Cycle 1 Week 15: number analyzed (eyes) | 134 | 134
  Cycle 1 Week 15 | 67.2 | 64.2
  Cycle 1 Week 20: number analyzed (Participants) | 10 | 10
  Cycle 1 Week 20: number analyzed (eyes) | 10 | 10
  Cycle 1 Week 20 | 50.0 | 40.0
  Cycle 1 Week 24: number analyzed (Participants) | 11 | 11
  Cycle 1 Week 24: number analyzed (eyes) | 11 | 11
  Cycle 1 Week 24 | 81.8 | 45.5
  Cycle 1 Week 28: number analyzed (Participants) | 11 | 11
  Cycle 1 Week 28: number analyzed (eyes) | 11 | 11
  Cycle 1 Week 28 | 63.6 | 45.5
  Cycle 1 Week 31: number analyzed (Participants) | 5 | 5
  Cycle 1 Week 31: number analyzed (eyes) | 5 | 5
  Cycle 1 Week 31 | 100.0 | 40.0
  Cycle 1 Week 36: number analyzed (Participants) | 11 | 11
  Cycle 1 Week 36: number analyzed (eyes) | 11 | 11
  Cycle 1 Week 36 | 72.7 | 72.7
  Cycle 1 Week 40: number analyzed (Participants) | 11 | 11
  Cycle 1 Week 40: number analyzed (eyes) | 11 | 11
  Cycle 1 Week 40 | 54.5 | 54.5
  Cycle 1 Week 44: number analyzed (Participants) | 11 | 11
  Cycle 1 Week 44: number analyzed (eyes) | 11 | 11
  Cycle 1 Week 44 | 81.8 | 45.5
  Cycle 1 Week 47: number analyzed (Participants) | 11 | 11
  Cycle 1 Week 47: number analyzed (eyes) | 11 | 11
  Cycle 1 Week 47 | 72.7 | 54.5
  Cycle 1 Week 52: number analyzed (Participants) | 11 | 11
  Cycle 1 Week 52: number analyzed (eyes) | 11 | 11
  Cycle 1 Week 52 | 81.8 | 81.8
  Cycle 2 Day 2: number analyzed (Participants) | 124 | 124
  Cycle 2 Day 2: number analyzed (eyes) | 124 | 124
  Cycle 2 Day 2 | 70.2 | 89.5
  Cycle 2 Week 4: number analyzed (Participants) | 125 | 125
  Cycle 2 Week 4: number analyzed (eyes) | 125 | 125
  Cycle 2 Week 4 | 68.8 | 75.2
  Cycle 2 Week 8: number analyzed (Participants) | 124 | 124
  Cycle 2 Week 8: number analyzed (eyes) | 124 | 124
  Cycle 2 Week 8 | 68.5 | 71.0
  Cycle 2 Week 12: number analyzed (Participants) | 118 | 118
  Cycle 2 Week 12: number analyzed (eyes) | 118 | 118
  Cycle 2 Week 12 | 72.0 | 65.3
  Cycle 2 Week 15: number analyzed (Participants) | 98 | 98
  Cycle 2 Week 15: number analyzed (eyes) | 98 | 98
  Cycle 2 Week 15 | 69.4 | 64.3
  Cycle 2 Week 20: number analyzed (Participants) | 91 | 91
  Cycle 2 Week 20: number analyzed (eyes) | 91 | 91
  Cycle 2 Week 20 | 76.9 | 64.8
  Cycle 2 Week 24: number analyzed (Participants) | 87 | 87
  Cycle 2 Week 24: number analyzed (eyes) | 87 | 87
  Cycle 2 Week 24 | 64.4 | 71.3
  Cycle 2 Week 28: number analyzed (Participants) | 85 | 85
  Cycle 2 Week 28: number analyzed (eyes) | 85 | 85
  Cycle 2 Week 28 | 76.5 | 74.1
  Cycle 2 Week 31: number analyzed (Participants) | 86 | 86
  Cycle 2 Week 31: number analyzed (eyes) | 86 | 86
  Cycle 2 Week 31 | 76.7 | 74.4
  Cycle 2 Week 36: number analyzed (Participants) | 91 | 91
  Cycle 2 Week 36: number analyzed (eyes) | 91 | 91
  Cycle 2 Week 36 | 79.1 | 67.0
  Cycle 3 Day 2: number analyzed (Participants) | 33 | 33
  Cycle 3 Day 2: number analyzed (eyes) | 33 | 33
  Cycle 3 Day 2 | 75.8 | 90.9
  Cycle 3 Week 4: number analyzed (Participants) | 31 | 31
  Cycle 3 Week 4: number analyzed (eyes) | 31 | 31
  Cycle 3 Week 4 | 74.2 | 71.0
  Cycle 3 Week 8: number analyzed (Participants) | 32 | 32
  Cycle 3 Week 8: number analyzed (eyes) | 32 | 32
  Cycle 3 Week 8 | 75.0 | 59.4
  Cycle 3 Week 15: number analyzed (Participants) | 30 | 30
  Cycle 3 Week 15: number analyzed (eyes) | 30 | 30
  Cycle 3 Week 15 | 70.0 | 43.3
  Cycle 3 Week 20: number analyzed (Participants) | 33 | 33
  Cycle 3 Week 20: number analyzed (eyes) | 33 | 33
  Cycle 3 Week 20 | 69.7 | 39.4

ADVERSE EVENTS:
Time Frame: First treatment to end of study (up to 525 days)
Description: All-cause Mortality: ITT Population included all randomized participants. Serious and Other AEs: Safety Population included all participants who received treatment and data is collected and presented as per randomization. Ocular AEs reported for Eye Disorders were collected for each eye (primary eye or contralateral eye) separately. The AE footnotes are used to report the number of AEs that occurred in the primary eye and in the contralateral eye. A participant could have ≥1 events.
Arm/Group | SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) | Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye)
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 11/72 | 6/70
Other Adverse Events (participants affected / at risk) | 56/72 | 44/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) (N=72) | Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) (N=70)
Myocardial infarction (Cardiac disorders) | 1 | 0
Corneal endothelial cell loss (Eye disorders) | 4 | 1 — 4 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=0, Contralateral Eye=4); 1 adverse event occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=1, Contralateral Eye=0).
Cataract (Eye disorders) | 1 | 0 — 1 adverse event occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=0, Contralateral Eye=1).
Corneal oedema (Eye disorders) | 0 | 2 — 2 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=2, Contralateral Eye=0).
Drug hypersensitivity (Immune system disorders) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Quadrantanopia (Nervous system disorders) | 1 | 0 — 1 adverse event occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=0, Contralateral Eye=1).
Dizziness (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal haematoma (Renal and urinary disorders) | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) (N=72) | Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) (N=70)
Conjunctival hyperaemia (Eye disorders) | 30 | 19 — 48 adverse events occurred in SLT (Primary Eye)/Bim SR 15 µg (Contralateral Eye) Arm:(Primary Eye=20,Contralateral Eye=28);27 adverse events occurred in Bim SR 15 µg(Primary Eye)/SLT (Contralateral Eye) Arm (Primary Eye=19, Contralateral Eye=8).
Corneal endothelial cell loss (Eye disorders) | 11 | 4 — 11 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=1, Contralateral Eye=10); 4 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=3, Contralateral Eye=1).
Punctate keratitis (Eye disorders) | 10 | 8 — 18 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=8, Contralateral Eye=10);14 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=8, Contralateral Eye=6).
Conjunctival haemorrhage (Eye disorders) | 7 | 5 — 8 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=1, Contralateral Eye=7); 7 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=5, Contralateral Eye=2).
Corneal oedema (Eye disorders) | 6 | 9 — 6 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=1, Contralateral Eye=5); 9 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=8, Contralateral Eye=1).
Photophobia (Eye disorders) | 6 | 4 — 8 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=2, Contralateral Eye=6); 6 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=4, Contralateral Eye=2).
Eye irritation (Eye disorders) | 6 | 3 — 10 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=4, Contralateral Eye=6); 5 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=3, Contralateral Eye=2).
Eye pain (Eye disorders) | 5 | 9 — 6 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=4, Contralateral Eye=2); 10 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=7, Contralateral Eye=3).
Dry eye (Eye disorders) | 5 | 3 — 8 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=4, Contralateral Eye=4); 4 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=3, Contralateral Eye=1).
Anterior chamber cell (Eye disorders) | 4 | 3 — 5 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=1, Contralateral Eye=4); 3 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=2, Contralateral Eye=1).
Foreign body sensation in eyes (Eye disorders) | 4 | 3 — 5 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=1, Contralateral Eye=4); 3 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=3, Contralateral Eye=0).
Corneal opacity (Eye disorders) | 4 | 0 — 4 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=1, Contralateral Eye=3).
Conjunctivitis (Infections and infestations) | 4 | 1 — 4 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=0, Contralateral Eye=4); 2 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=1, Contralateral Eye=1).
Sinusitis (Infections and infestations) | 1 | 4
Intraocular pressure increased (Investigations) | 13 | 7 — 18 adverse events occurred in SLT (Primary Eye) / Bim SR 15 µg (Contralateral Eye) Arm: (Primary Eye=8, Contralateral Eye=10);12 adverse events occurred in Bim SR 15 µg (Primary Eye) / SLT (Contralateral Eye) Arm (Primary Eye=6, Contralateral Eye=6).
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4
Headache (Nervous system disorders) | 3 | 4
Hypertension (Vascular disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT02636946/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT02636946/SAP_001.pdf